CLINICAL TRIAL: NCT03989427
Title: The Effectiveness of Brushing and Flossing Sequence on Control of Plaque and Gingival Inflammation-A Randomized Controlled Clinical Trial in Klinik Pergigian, MMMC, Melaka
Brief Title: The Effectiveness of Brushing and Flossing Sequence on Control of Plaque and Gingival Inflammation
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melaka Manipal Medical College (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Principal Investigator, Rajesh Hosadurga, Professor, Melaka Manipal Medical College
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: MMMC/FOD/AR/B6
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Gingival Inflammation; Plaque; Gingival Bleeding; Plaque Control
Keywords: Gingiva; Gingivitis; Flossing; Brushing; Plaque control; Gingival bleeding; Bleeding point index; Rustogi Modified Navy Plaque Index; Dental Plaque; Tooth brushing
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid; Gingival Hemorrhage; Dental Plaque

STUDY DESIGN:
Intervention Model Description: Participants will be selected by random sampling and allocated to Two Arms: Arm-I - Brushing first and Flossing later (BF), Arm II- Flossing first and brushing later (FB) after applying inclusion and exclusion criteria.
  The participants in BF group will Brush first using Colgate® tooth brush for a 2-week period. and then floss with Colgate® dental floss using Spool method for a 2-week period. This is followed by a one week wash out period After this cross over is done in which participants will change the sequence to FB wherein they will floss first and brush later.
  The participants in FB group will floss first with Colgate® dental floss and brush later using Colgate® tooth brush for a 2-week period. This is followed by a one week wash out period. After this cross over is done in which participants will change the sequence to BF wherein they will Brush first and Floss later.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will record measurements at baseline and post intervention. The assessor will be blinded from the sequence of intervention allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brushing First and Flossing Later (BF) (Experimental): The participants in BF group were asked to use modified bass method of tooth brushing first using Colgate® tooth brush (the amount of Colgate® tooth paste used is half-length of the toothbrush's head) and then floss with Colgate® dental floss using Spool method for a 2-week period. This is followed by a one week wash out period wherein they will practice oral hygiene according to their habitual method. After this cross over is done in which participants will change the sequence to FB wherein they will floss first and brush later.
  Interventions: Other: Brushing first and Flossing later (BF)
- Flossing First and Brushing Later (FB) (Experimental): The participants in FB group were asked to floss first with Colgate® dental floss using Spool method and then modified bass method of tooth brushing first using Colgate® tooth brush (the amount of Colgate® tooth paste used is half-length of the toothbrush's head) for a 2-week period. This is followed by a one week wash out period wherein they will practice oral hygiene according to their habitual method. After this cross over is done in which participants will change the sequence to BF wherein they will brush first and floss later.
  Interventions: Other: Flossing first and Brushing later (FB)

INTERVENTIONS:
Other: Brushing first and Flossing later (BF) — Participants will follow Brushing first and flossing later (BF) sequence for 2 weeks, and after 1 week wash out period, Flossing first and Brushing later (FB) sequence for another 2 weeks.
  Other Names: Colgate® tooth brush and Colgate® Dental Floss
  Arms: Brushing First and Flossing Later (BF)
Other: Flossing first and Brushing later (FB) — Participants will follow Flossing first and Brushing later (FB) sequence for 2 weeks, and after 1 week wash out period, Brushing first and flossing later (BF) sequence for another 2 weeks.
  Other Names: Colgate® tooth brush and Colgate® Dental Floss
  Arms: Flossing First and Brushing Later (FB)

SUMMARY:
This study evaluates the effectiveness of brushing and flossing sequence in the control of dental plaque and gingival inflammation.

DETAILED DESCRIPTION:
Periodontal disease is the disease of the supporting dental tissues like alveolar bone,periodontal ligament cementum and gingiva. The most common form is plaque-induced gingivitis . Bleeding on gingival probing is one of the hallmarks of gingival inflammation.The removal of dental plaque is the most crucial action for preventing and treating gingival inflammation. Toothbrush along with toothpaste are still the most reliable means of plaque control. However, cleaning should be thorough and performed at regular intervals.

Toothbrush has a limited ability to reach all the areas around the tooth. Inter-dental areas are prone for plaque accumulation and gingival inflammation. Dental floss is one of the most effective tool in addition to tooth brush to remove inter-dental plaque. The sequence of using toothbrush and dental floss may influence the removal of dental plaque and consequently reducing the bleeding on probing of gingiva. There is conflicting evidence in the literature. The hypothesis of this study is that the sequence of brushing and flossing will not influence control of plaque control and gingival inflammation.

ELIGIBILITY:
Inclusion Criteria:

• Dental students of Dental school of Melaka-Manipal Medical College

Exclusion Criteria:

* Participants who had systemic diseases
* Gingivitis or periodontitis
* Use of antibiotics in the past 3 months,
* Pregnancy,
* Smoking
* Orthodontic appliances.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Rashid Ismail, BDS, Study Director — Melaka Manipal Medical College
Locations (1):
- Faculty of Dentistry, Melaka-Manipal Medical College, Melaka Tengah, Melaka, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
If Requested by authors for systematic review, study results will be shared for secondary research.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January 2020- January 2023
Access Criteria: IPD access will be given only to bona fide research groups as evidenced via their resume and the involvement of a qualified statistician.
  Consent will be taken from the participants about data sharing prior to the commencement of the study. Confidentiality will be strictly maintained.
  Data custodians are scientific committee, Faculty of Dentistry, MMMC, Melaka. Data access will be reviewed and approved by DRC based on Merits of requests.

REFERENCES:
- [Background] Torkzaban P, Arabi SR, Sabounchi SS, Roshanaei G. The Efficacy of Brushing and Flossing Sequence on Control of Plaque and Gingival Inflammation. Oral Health Prev Dent. 2015;13(3):267-73. doi: 10.3290/j.ohpd.a32678. PMID 25197738
- [Background] Mazhari F, Boskabady M, Moeintaghavi A, Habibi A. The effect of toothbrushing and flossing sequence on interdental plaque reduction and fluoride retention: A randomized controlled clinical trial. J Periodontol. 2018 Jul;89(7):824-832. doi: 10.1002/JPER.17-0149. Epub 2018 Jul 20. PMID 29741239
- [Background] Zanatta FB, Antoniazzi RP, Pinto TM, Rosing CK. Supragingival plaque removal with and without dentifrice: a randomized controlled clinical trial. Braz Dent J. 2012;23(3):235-40. doi: 10.1590/s0103-64402012000300009. PMID 22814692
- [Background] Valkenburg C, Slot DE, Bakker EW, Van der Weijden FA. Does dentifrice use help to remove plaque? A systematic review. J Clin Periodontol. 2016 Dec;43(12):1050-1058. doi: 10.1111/jcpe.12615. Epub 2016 Oct 3. PMID 27513809
- [Background] Jayakumar A, Padmini H, Haritha A, Reddy KP. Role of dentifrice in plaque removal: a clinical trial. Indian J Dent Res. 2010 Apr-Jun;21(2):213-7. doi: 10.4103/0970-9290.66629. PMID 20657090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 221 students were screened for eligibility between January 25, 2019 to May 10, 2019 in the Out-Patient Department (OPD) of Dept.of Periodontics, Poly clinic A, Klinik Pergigian, Melaka, Malaysia.
Pre-assignment Details: 30 of 221 participants were randomized. Of those not randomized, 120 did not meet inclusion criteria and 71 declined to participate.
Groups:
- Brushing Flossing (BF): Participants used Brushing first and Flossing (BF) sequence in the study. After 1 week wash out period they used Flossing first and brushing (FB) later sequence.
  Toothbrush used was Colgate® tooth brush- Soft bristled, waxed dental floss (Colgate® dental floss) and toothpaste (Colgate® tooth paste) were standardized.
  The method of brushing used was Modified Bass Method, the amount of dentifrice used is half-length of the toothbrush's head and Spool method of flossing was used.
- Flossing Brushing (FB): Participants used Flossing first and brush (FB) later sequence in the study. After 1 week wash out period they used Brushing first and flossing (FB) later sequence.
  Toothbrush used was Colgate® tooth brush- Soft bristled, waxed dental floss (Colgate® dental floss) and toothpaste (Colgate® tooth paste) were standardized.
  The method of brushing used was Modified Bass Method, the amount of dentifrice used is half-length of the toothbrush's head and Spool method of flossing was used.
Period: First Intervention (2 Weeks)
Arm/Group | Brushing Flossing (BF) | Flossing Brushing (FB)
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Brushing Flossing (BF) | Flossing Brushing (FB)
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | Brushing Flossing (BF) | Flossing Brushing (FB)
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Brushing Flossing (BF) First: Participants used Brushing first and Flossing later (BF) sequence for 2 weeks. After a washout period of 1 week they used flossing first and brushing later (FB) sequence
  Toothbrush used was Colgate® tooth brush- Soft bristled, waxed dental floss (Colgate® dental floss) and toothpaste (Colgate® tooth paste) were standardized.
  The method of brushing used was Modified Bass Method, the amount of dentifrice used is half-length of the toothbrush's head. The method of flossing used was Spool method of flossing.
- Flossing Brushing (FB) First: Participants used Flossing first and Brushing later (FB) sequence for a period of 2 weeks. After a washout period of 1 week they used Brushing first and flossing later (BF) sequence
  Toothbrush used was Colgate® tooth brush- Soft bristled, waxed dental floss (Colgate® dental floss) and toothpaste (Colgate® tooth paste) were standardized.
  The method of brushing used was Modified Bass Method, the amount of dentifrice used is half-length of the toothbrush's head and the method of flossing used was Spool method of flossing.
- Total: Total of all reporting groups
Arm/Group | Brushing Flossing (BF) First | Flossing Brushing (FB) First | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.87 (0.52) | 23.00 (0.38) | 22.93 (0.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 1 | 3 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Malaysian Malay | 6 | 6 | 12
  Malaysian Chinese | 3 | 4 | 7
  Malaysian Indians | 4 | 3 | 7
  others | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Malaysia | 15 | 15 | 30
BPI scores [Mean (Standard Deviation); unit: units on a scale] — Bleeding on probing will determined at the buccal, lingual and proximal surfaces using the Changes in BPI (Bleeding on probing index ) scores will be used to assess change in bleeding on probing scores at baseline and end of the 1st phase of the study( where the participants will brush first and then floss) and at the end of the 2nd phase (where the participants will floss first and brush later).
  BPI score- minimum value is 0% and Maximum is 100% of bleeding surfaces. Higher mean score is poor outcome.
  However, higher reduction in mean score compared to baseline is better outcome.
  units on a scale | 1.8840 (1.765) | 2.5253 (2.388) | 2.2047 (2.089)
RMNPI index scores [Mean (Standard Deviation); unit: units on a scale] — Rustogi Modified Navy Plaque Index(RMNPI) is used to assess change in plaque scores at baseline. Maximum number of surfaces examined are 504. Minimum value is 0 and maximum value is 1 in each patient.
  The measure of dispersion used was Mean and Standard error. A positive error means that the predicted value is larger than the true value, and a negative error means that the predicted value is less than true value. The mean error should be close to zero. Higher mean score is a worse outcome.Higher percent reduction in mean score when compared to baseline is better outcome.
  units on a scale | 0.0866 (0.687) | 0.025 (0.020) | 0.080 (0.066)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean BPI Index Scores at 2 Weeks
Description: Bleeding on probing (BOP) is an objective indicator of inflammation. BPI (Bleeding Point Index) is a validated index used to measure BOP. BOP is determined at the buccal, lingual and proximal surfaces of all teeth using BPI scores. BPI scores are measured at baseline and 2 weeks, followed by a wash out period of one week. BPI score is measured again at baseline and 2 weeks after cross over in intervention. Change in BPI scores will give the estimation of effect of the intervention. BPI score- minimum value is 0% and Maximum is 100% of bleeding surfaces in each individual patient with teeth. A positive error means that the predicted value is larger than the true value, and a negative error means that the predicted value is less than the true value. The mean error should be close to zero. Sometimes it will be negative or positive depending on the population.. Higher mean score is poor outcome. However, higher reduction in mean score compared to baseline is better outcome.
Time Frame: Baseline and 2 weeks
Population: All participants who received at least one intervention each and completed all study visits were included in the effectiveness analysis.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Brushing First and Flossing Later (BF): Participants who performed Brushing first and flossing later (BF) in either the first or last 2 weeks of the study
- Flossing First and Brushing Later (FB): Participants who performed Flossing first and brushing later (FB) in either the first or last 2 weeks of the study.
Arm/Group | Brushing First and Flossing Later (BF) | Flossing First and Brushing Later (FB)
Number analyzed (Participants) | 30 | 30
score on a scale | 0.396 (0.410) | -1.028 (0.392)
Statistical Analysis 1: Comparison: Brushing First and Flossing Later (BF) vs Flossing First and Brushing Later (FB); Null hypothesis is that the sequence of brushing first and flossing later has no effect on gingival inflammation. No previous studies with Mean and SD were available. Hence, a pilot study was done. 30 participants were randomly assigned to Brush first and floss later (BF) group ; and Floss first brush later(FB) group. After 1 week there was cross-over. 80% power is required to detect mean difference in BPI scores; Test type: Equivalence — The two treatment sequence could be called equivalent if the observed difference and its 95% CI are completely inside the interval of clinical equivalence. A significant result (p < 0.05) means that the two treatments are equivalent, according the definition of equivalence as defined clinically; p = 0.022, ANOVA — The threshold for statistical significance was p <0.05; Three-way mixed ANOVA was done to determine the effect of Intervention on BPI scores; Mean Difference (Net) = 1.424, 95% CI 2-sided [0.221 to 2.628]

2. Secondary Outcome: Change From Baseline in Mean RMNPI Index Score at 2 Weeks
Description: Rustogi Modified Navy Plaque Index(RMNPI) is a self validated tool to assess dental plaque accumulation on the teeth surfaces. RMNPI scores are used to assess change in plaque scores at baseline and at the end of 2 weeks .This will be followed by a 1 week wash out period. Then there is a cross over in the intervention. RMNPI scores are measured again from Baseline and 2 weeks. Maximum number of surfaces examined are 504 per person. A Minimum value of 0 and maximum value of 1 can be calculated in each patient.
  Higher mean score is a worse outcome. However,higher percent reduction in mean score when compared to baseline is better outcome.
Time Frame: Baseline and 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Brushing First and Flossing Later (BF): Participants who performed Brushing First and Flossing Later(BF) in either the first or last 2 weeks of the study.
Arm/Group | Brushing First and Flossing Later (BF) | Flossing First and Brushing Later (FB)
Number analyzed (Participants) | 30 | 30
score on a scale | 0.042 (1.043) | 0.101 (1.427)
Statistical Analysis 1: Comparison: Brushing First and Flossing Later (BF) vs Flossing First and Brushing Later (FB); Null hypothesis: The sequence of brushing and flossing has no effect on plaque scores There were no previous studies with Mean and SD to calculate sample. So a pilot study was conducted. 30 participants were randomly assigned in 1:1 fashion to Brush-floss (GroupA) and Floss brush group (group B). Then after 1 week there was cross-over among the groups.2 groups would have at least 80% power to detect the mean difference in BPI scores; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.971, ANOVA; Three-way mixed ANOVA was done to determine the effect of Intervention on RMNPI index scores; Mean Difference (Net) = -0.058, 95% CI 2-sided [-3.335 to 3.219]

ADVERSE EVENTS:
Time Frame: Baseline, 24 hours, 2 weeks, 5 weeks
Description: We followed the description provided by clinical trials. gov. Adverse event and serious adverse event was recorded in our data collection sheet for each participant. Checklist was prepared for each participant and attached to the data form. The data was recorded at baseline examination carried out in the morning clinical session, the participants were reviewed after 24 hours, 2 weeks and 5 weeks. They were asked to report immediately if any adverse events occurred in other periods of time.
Groups:
- Brushing and Flossing: No adverse events were reported
Arm/Group | Brushing and Flossing
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
There was no article with available to calculate sample size. Hence we conducted the pilot study among 30 participants. We recalculated the sample size from mean and SE of our study. It was estimated to be 40.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT03989427/Prot_000.pdf
  • Informed Consent Form (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT03989427/ICF_001.pdf
  • Statistical Analysis Plan (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT03989427/SAP_002.pdf